CLINICAL TRIAL: NCT01746823
Title: Identification of Disease Progression Specific Biomarkers and Their Pharmacologic Modulation for Keratoconus.
Brief Title: Identification and Validation of Functional Biomarkers for Keratoconus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Narayana Nethralaya (Other)
Collaborators: Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, Dr Rohit Shetty, Consultant, Cornea and Refractive Services, Narayana Nethralaya
Other Study IDs: NNKC-2011
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2012-12

CONDITIONS: Keratoconus
Keywords: Keratoconus; Proteomics
MeSH Terms: conditions — Keratoconus | interventions — Cyclosporins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Tear samples and discarded epithelium from Keratoplasty surgeries.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Controls, Keratoconus: Sub group of Keratoconus to be treated with anti-inflammatory agents ie Cyclosporine-A
  Interventions: Drug: Cyclosporins

INTERVENTIONS:
Drug: Cyclosporins
  Other Names: Restasis

SUMMARY:
There is currently no medication for containing KC, nor any adequate biomarkers to predict the disease. Furthermore, there is considerable confusion in the field regarding the pathophysiology of the disease and involvement of inflammation. To that end, this study is designed to address some of these questions by determining the proteomic profiles of KC patients with different clinical grades. This relatively large cohort study is expected to yield significant information regarding the molecules that are deregulated during progression of KC and may provide a framework to assign diagnostic biomarkers and therapeutic intervention points.

DETAILED DESCRIPTION:
The screening of keratoconus involves keratoconus related clinical signs like retinoscopy scissors reflex, Munson sign, stromal thinning, Vogt's striae, and Fleischer's ring, but corneal topography is the most useful method in the diagnosis of keratoconus, especially in the absence of clinical signs.

Several devices are currently available for detecting early keratoconus by measuring anterior and posterior corneal topography and elevation(Mihaltz et al. 2009; Ishii et al. 2012). Corneal topographic and tomographic techniques which generate color-coded maps and topographic indices, are the most sensitive devices for confirming the diagnosis of keratoconus(Rabinowitz 1998; Rao et al. 2002) were used for diagnosis in this study. In addition, videokeratography has been shown to identify Forme fruste keratoconus (FFKC) in the absence of clinical signs of keratoconus. Videokeratographic indices such as the Klyce/Maeda criteria, the Rabinowitz criteria, and others have been developed to quantitatively analyze videokeratography and screen for keratoconus(Rao et al. 2002). These indices have been shown to identify keratoconus with a high degree of sensitivity and specificity. The Orbscan II is a three-dimensional slit-scan topography system for analysis of the corneal surfaces and anterior chamber and has been used on all patients in the study. It uses calibrated video and a scanning slit beam to measure x, y, and z locations of several thousand points. These points are used to construct topographic maps(Rao et al. 2002). The Pentacam (Oculus Inc) is a corneal tomographer technology which generates data on topograophy and elevation of anterior and posterior using a rotating Scheimpflug camera which has also been used on all subjects enrolled in this study. Various diagnostic parameters are available for keratoconus diagnosis depending on what mode of topography is being used. Maeda and Klyce designed a system to detect keratoconus. The system, which is based on linear discriminant analysis and a binary decision tree, identifies the map as representing keratoconus or nonkeratoconus and, based on a value from the discriminant analysis (the KPI), assigns the map an index expressed as a percentage that suggests the severity of keratoconus. At this time, however, Keratoconus Severity Index (KSI) and the Amsler-Krumeich classification are the most popular methods for grading keratoconus severity(Mihaltz et al. 2009; Ishii et al. 2012). KSI is based on indices estimated by a curvature map using Placido disk-based corneal topography, and Amsler-Krumeich classification defines the stage of keratoconus using biomicroscopy, mean central keratometry reading, spherical and cylindrical refraction change, and corneal thickness(Mihaltz et al. 2009; Ishii et al. 2012). This is the index that has been used for the final gradation of keratoconus stages of all subjects in this study.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of corneal thinning by any type of keratometry

Exclusion Criteria:

* Corneal inflammation without evidence of ectasia
* Retinal disorder subjects excluded

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients detected with corneal thinning by keratometry at a tertiary level hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Keratoconus grade specific biomarker identification | 1 year

SECONDARY OUTCOMES:
Onlabel use of anti-allergic topical treatment for inhibition of specific biomarkers to modify keratoconus disease progression | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Shetty, MBBS,DNB, FRCS, Principal Investigator — Narayana Nethralaya
Locations (1):
- Narayana Nethralaya, Bangalore, Karnataka, India

REFERENCES:
- [Background] Gontier J, Fisch U. Schirmer's test: its normal values and clinical significance. ORL J Otorhinolaryngol Relat Spec. 1976;38(1):1-10. doi: 10.1159/000275252. PMID 943747
- [Derived] Shetty R, Ghosh A, Lim RR, Subramani M, Mihir K, Reshma AR, Ranganath A, Nagaraj S, Nuijts RM, Beuerman R, Shetty R, Das D, Chaurasia SS, Sinha-Roy A, Ghosh A. Elevated expression of matrix metalloproteinase-9 and inflammatory cytokines in keratoconus patients is inhibited by cyclosporine A. Invest Ophthalmol Vis Sci. 2015 Feb 3;56(2):738-50. doi: 10.1167/iovs.14-14831. PMID 25648341